CLINICAL TRIAL: NCT00838357
Title: Plerixafor and G-CSF for the Mobilisation of Peripheral Blood Stem Cells for Autologous Stem Cell Transplantation in Patients With Non-Hodgkin's Lymphoma (NHL), Hodgkin's Disease (HD) or Multiple Myeloma (MM) - Safety Study in a General Autologous Transplant Population
Brief Title: A Multi-centre, Open Label, Single-arm Study Intended to Further Investigate the Safety and Efficacy of Plerixafor as a Front-line Mobilisation Agent in Combination With G-CSF in Patients With Lymphoma or MM (Multiple Myeloma).
Acronym: PREDICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOZ00808; 2008-000689-21 (EudraCT Number)
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma (Non-Hodgkin's Lymphoma); Hodgkin's Disease or Multiple Myeloma; Front Line Mobilization; Transplantation
Keywords: Mobilisation stem cells; G-CSF Mobilisation Regimen; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor (Experimental): Plerixafor added to a G-CSF Mobilisation regimen
  Interventions: Drug: Generic = Plerixafor

INTERVENTIONS:
Drug: Generic = Plerixafor — 240µg/kg administered as an SC injection 10 to 11 hours prior to initiation of apheresis. Daily administration for 1 up to 5 consecutive days

SUMMARY:
This is a research study intended to further investigate the safety and efficacy of plerixafor in patients with NHL, HD, or MM. Patients who have previously failed stem cell mobilisation attempts or who have previously received more than one autologous or any allogeneic stem cell transplant are not eligible.

DETAILED DESCRIPTION:
Patients with advanced or treatment-refractory Multiple Myeloma (MM), Hodgkin's Disease (HD) and Non-Hodgkin's Lymphoma (NHL) may be successfully treated with high dose chemotherapy followed by autologous transplantation of peripheral blood stem cells (PBSCs). Successful engraftment of peripheral blood stem cells (PBSCs) is well correlated with the number of CD34+ cells infused.

Stem cell collection with plerixafor could have a major benefit by increasing the circulating number of PBSCs and decreasing the number of apheresis sessions required to collect a sufficient number of PBSCs for transplant.

This is a multi-centre, open label, single-arm study intended to further investigate the safety and efficacy of plerixafor in patients with NHL, HD, or MM. Patients who have previously failed stem cell mobilisation attempts or who have previously received more than one autologous or any allogeneic stem cell transplant are not eligible.

Screening for eligibility will take place up to 30 days before the first dose of G-CSF. Patients will receive a stem cell mobilisation regimen consisting of plerixafor and G-CSF. Patients will be given G-CSF for 4 consecutive days in the morning. Starting on the evening of Day 4, plerixafor will be administered subcutaneously (SC). The plerixafor dose will be timed to allow for a 10- to 11-hour interval between the plerixafor dosing and the initiation of apheresis. Patients may continue to receive the evening dose of plerixafor then G-CSF the next morning followed by apheresis for up to a total of 5 apheresis procedures until a minimum of at least 5 x 106 CD34+ cells/kg for NHL/HD or 6 x 106 CD34+ cells/kg for MM are collected. More cells may be collected if done within the 5 apheresis procedures. Stem cell collection will take place using standard procedures.

Following the last apheresis, patients will undergo pre-transplant myeloablative chemotherapy followed by transplantation of the collected autologous stem cells, using the established protocols and procedures at each site.

Peripheral blood samples will be collected for determining the number of CD34+ cells in the peripheral blood. In addition, a sample will be obtained from each apheresis product to determine the quantity of CD34+ cells collected after each procedure.

Safety data will be reported according to guidelines provided in the protocol. Adverse event (AE) guidance is summarised in the protocol. Investigators will grade AEs using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.

Efficacy will be based on the quantity of CD34+ cells harvested and the subsequent engraftment and graft status. Patients who undergo haematopoietic stem cell transplantation will be monitored for graft status at 100 days, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM, NHL, or HD in partial response (PR) or complete response (CR)
* Eligible and planned for an autologous haematopoietic stem cell transplantation
* Written informed consent
* At least 18 years of age (inclusive)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* White blood cell (WBC) count ≥2.5 x 10^9/L
* Absolute neutrophil count (ANC) ≥1.5 x 10^9 /L
* Platelet count ≥100 x 10^9/L
* Serum creatinine ≤2.2 mg/dL
* Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT), and total bilirubin <2.5 x upper limit of normal (ULN)
* Adequate cardiac, renal, and pulmonary function sufficient to undergo apheresis and transplantation, i.e., eligible by institutional standards for autologous stem cell transplant
* All patients must agree to use a highly effective method of contraception whilst on study treatment and for at least 3 months following plerixafor treatment (including both female patients of child-bearing potential and male patients with partners of child-bearing potential). Effective birth control includes: a) birth control pills, depot progesterone, or an intrauterine device plus one barrier method, or b) two barrier methods. Effective barrier methods are: male and female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). For patients using a hormonal contraceptive method, information about any interaction of plerixafor with hormonal contraceptives is not known.

Exclusion Criteria:

* History of any acute or chronic leukaemia (including myelodysplastic syndrome)
* Prior allogeneic transplantation or more than one prior autologous transplantation
* Failed previous CD34+ cell collection attempts (either due to insufficient yield in apheresis product, or ineligible for apheresis because of inadequate mobilisation of CD34+ cells into peripheral blood)
* Less than 4 weeks since last anti-cancer therapy (including chemotherapy, biologic/immunologic, radiation) or less than 6 weeks if prior therapy with nitrosourea or mitomycin (for therapies with long-acting agents, a treatment-free interval of at least 2 half-lives should be considered) with the exception of ; Treatment with thalidomide, dexamethasone, lenalidomide (Revlimid®), and/or bortezomib (Velcade®) which is allowed up to 7 days prior to the first dose of G-CSF.
* Bone marrow involvement >20% assessed based on the most recent bone marrow aspirate or biopsy
* Treated with G-CSF or other cytokine within 14 days prior to the first dose of G-CSF for mobilisation
* Known to be human immunodeficiency virus (HIV) positive
* Active hepatitis B or hepatitis C
* Acute infection (febrile, i.e., temperature >38°C) within 24 hours prior to dosing or antibiotic therapy within 7 days prior to the first dose of G-CSF
* Hypercalcaemia as evidenced by >1 mg/dL above ULN
* Previously received investigational therapy within 4 weeks of enrolling in this protocol or currently enrolled in another investigational protocol during the mobilisation phase
* Central nervous system involvement including brain metastases or leptomeningeal disease
* Pregnant or nursing women
* Electrocardiogram (ECG) or study result (exercise study, scan) indicative of cardiac ischaemia or a history of clinically significant rhythm disturbance (arrhythmias), or other conduction abnormality in the last year that in the opinion of the Investigator warrants exclusion of the subject from the trial.
* Co-morbid condition(s), which in the opinion of the Investigator, renders the patient at high risk from treatment complications or impairs their ability to comply with the study treatment and protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To confirm the safety profile of plerixafor to mobilise stem cells when used in patients with lymphoma or MM who are eligible to undergo treatment with an autologous haematopoietic stem cell transplant | 24 months

SECONDARY OUTCOMES:
To assess efficacy of plerixafor and granulocyte-colony stimulating factor (G-CSF) as a mobilisation regimen as measured by the number of CD34+ cells collected in each apheresis session | After each dose of plerixafor
To assess the clinical effectiveness of plerixafor and G-CSF mobilised stem cells by examining haematopoietic cell engraftment and graft status | After transplantation
To examine the influence of CD34+ cell dose infused on time to engraftment, engraftment and graft status | After transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Europe B.V.
Locations (26):
- France (6):
  - Hôpital du Haut Lévêque, Bordeaux
  - Hôpital Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Hotel-Dieu Université de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Charité - Campus Benjamin Franklin, Berlin
  - Klinikum der Universität zu Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitätsklinik Würzburg, Würzburg
- Italy (3):
  - L. & A. Seragnoli, University of Bologna, Bologna
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera S. Martino, Genova
- VU Medisch Centrum, Amsterdam, Netherlands
- Spain (4):
  - Hospital Santa Creu y Sant Pau, Barcelona
  - Hospital Carlos-Haya, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital la Fe, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (4):
  - Gartnavel Hospital, Glasgow
  - St James's University Hospital, Leeds
  - King's college Hospital, London
  - Nottingham University NHS Trust, Nottingham